CLINICAL TRIAL: NCT06972745
Title: Cohort Study on Efficacy and Tolerance of Right Unilateral Electroconvulsive Therapy vs. Bitemporal in Patients With Paranoid Schizophrenia in Acute Psychosis at Fray Bernardino Álvarez Psychiatric Hospital
Brief Title: Efficacy & Tolerability of Rigth Unilateral vs. Bitemporal ECT in Schizophrenia in a Psychiatric Hospital in Mexico
Acronym: ULTEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in operative and administrative functions
Sponsor: Hospital Psiquiátrico Fray Bernardino Álvarez (Other)
Responsible Party: Principal Investigator, Héctor Octavio Castañeda González, Attending Psychiatrist, Psychiatric Emergency Department, Hospital Psiquiátrico Fray Bernardino Álvarez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-962
Record Dates: First submitted 2025-04-20; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia Disorders
Keywords: Electroconvulsive teraphy; Schizophrenia; Rigth unilateral; Cognition; Efficacy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rigth unilateral electrode placement (Experimental): Anode (Right Temporal): Centered over the right temporal lobe, 2.5 cm (1 inch) above the midpoint of an imaginary line connecting the tragus and the external canthus.
  Cathode (Right Parietal): Placed vertically 10 cm (4 inches) above the temporal electrode, aligned with the parietal bone (midline between the temporal and occipital regions).
  Interventions: Procedure: Ultrabrief pulse electroconvulsive therapy
- Bitemporal electrode placement (Active Comparator): Anode placed over the left temporal region: Positioned 2.5 cm (1 inch) above the midpoint of an imaginary line connecting the tragus (ear canal) and the external canthus (outer corner) of the left eye.
  Catode positioned over the right temporal region: Mirror placement on the right side, symmetrically aligned with the left electrode.
  Interventions: Procedure: Brief pulse Electroconvulsive therapy

INTERVENTIONS:
Procedure: Ultrabrief pulse electroconvulsive therapy — Therapeutic seizure induction with pulse unidirectional electric charge through the right hemisphere, using ultrabrief pulses (≤0.3 ms).
  Arms: Rigth unilateral electrode placement
Procedure: Brief pulse Electroconvulsive therapy — Therapeutic seizure induction with pulse unidirectional electric charge through the temporal hemisferes, using brief pulses (≥0.5 ms).
  Arms: Bitemporal electrode placement

SUMMARY:
Electroconvulsive therapy (ECT) is an established treatment for medication-resistant schizophrenia. There is debate about the best method of electrode placement. Bitemporal (BT) placement is commonly used for schizophrenia, while right unilateral (RUL) placement in mood disorders is associated with fewer adverse effects on memory and language. This study compares the efficacy, safety and cognitive effects of BT-ECT versus RUL-ECT in hospitalized schizophrenia patients with acute psychosis.

Main Question: Does RUL-ECT reduce psychotic symptoms with fewer cognitive effects versus BT-ECT in patients with severe schizophrenia? Hypothesis: RUL-ECT is as effective as BT-ECT in reducing psychotic symptoms with fewer cognitive effects.

Methods: Randomized trial in patients with schizophrenia (confirmed by DSM 5 criteria) and severe symptoms (PANSS score ≥60). Patients were assigned to receive BT-ECT or RUL-ECT. Efficacy was measured by a ≥30% reduction in symptom severity on the PANSS scale and overall improvement measured with the Clinical Global Impression scale. Cognitive function was assessed with the Montreal Cognitive Assessment (MoCA) and Brief Assessment of Cognition in Schizophrenia (BACS) scales.

DETAILED DESCRIPTION:
Study Design and Setting: Randomized experimental trial at Fray Bernardino Álvarez Psychiatric Hospital, Mexico City.

Sample Size: Quota sampling. Eligibility Criteria: inpatients, spanish-speaking, ≥18 years old with DSM-5 schizophrenia diagnosis, PANSS total score ≥60, and treatment with 1-2 antipsychotics (including clozapine). Exclusions: ECT within 3 months, affective comorbidities, catatonia, pregnancy, anesthesia/ECT contraindications, or incomplete follow-up.

Equipment and Technique: Pre-ECT evaluations included ECG, chest X-ray, blood tests, and assessments by internists/anesthesiologists. ECT was administered by a principal investigator (Emory University-certified) using a MECTA Corp spECTrum 5000Q device, 3x/week (excluding weekends). Electrode placement: bitemporal (BT) with brief pulses (≥0.5 ms) or right unilateral (RUL; D'Elia placement) with ultrabrief pulses (≤0.3 ms). Initial titration doses: 48 mC (BT) or 4.8 mC (RUL), doubled until adequate seizure (assessed via Clinical and Seizure Based Stimulation method). Maintenance doses: 2x threshold (BT) or 6x threshold (RUL), adjusted by 50% for poor-quality seizures. Premedication: atropine (1 mg IM), propofol (1 mg/kg IV), and succinylcholine (1 mg/kg IV).

Intervention and Comparator: Active comparator: BT-ECT vs. RUL-ECT.(intervention) No placebo group due to institutional constraints.

Randomization and Blinding: Block randomization (Microsoft Excel-generated) by an independent researcher. Allocation sequence concealed by an assistant and disclosed pre-treatment.

Outcomes: Efficacy: ≥30% PANSS reduction; Safety: Adverse event frequency/severity/time to adverse event onset. Cognition: MoCA and BACS pre-/post-ECT (administered by neuropsychology-trained staff).

Ethics: Conducted per WMA Declaration of Helsinki. Informed consent obtained from patients' legal guardians due to severe mental impairment in participants

ELIGIBILITY:
A) Inclusion Criteria:

1. Spanish-speaking.
2. any sex/gender.
3. Aged ≥18 years.

3. Diagnosis of schizophrenia per DSM-5 criteria. 4. Baseline PANSS (Positive and Negative Syndrome Scale) total score ≥60. 5. Treatment with 1-2 antipsychotics (including clozapine).

B)Exclusion Criteria:

1. Received ECT (electroconvulsive therapy) within the previous 3 months.
2. Comorbid affective disorders (e.g., bipolar disorder, major depressive disorder).
3. Catatonia or catatonic syndrome.
4. Pregnancy
5. Contraindications to general anesthesia/ECT (i.e. uncontrolled cardiovascular disease or intracranial hypertension).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Efficacy of electroconvulsive therapy technique | 48 hours after last ECT session
  Treatment response is defined as a ≥20% reduction in the total score of the Positive and Negative Syndrome Scale (PANSS) after treatment. A dichotomous classification was applied (responders vs. non-responders) The PANSS assesses symptom severity through 30 items, each scored on a 1-7 scale, where: 1 = Absent (no symptom) and 7 = Extreme (severe symptom). Higher PANSS scores indicate greater symptom severity, meaning a lower score reflects a better clinical outcome.

SECONDARY OUTCOMES:
Adverse effect incidence | Between two hours and 24 hours after the last ECT session
  The incidence of side effects will be expressed as the percentage of subjects affected within each study group.
Time to adverse event onset measured in number of sessions | From the first session until 48 hours after last session
  Time to adverse event onset is defined as the number of completed ECT sessions where the outcome is first documented. Count of sessions from Session 1 (baseline) to the session where the AE is first documented.
Cognitive changes measured by MoCA | 48 hours after last ECT session
  Change in total Montreal Cognitive Assessment (MoCA) score at the end of treatment. Result will be analyzed as a continuous linear variable.
  MoCA evaluates 7 domains, with item-level binary scoring (0/1). Serial-7s allow up to 3 points (1 per correct subtraction). Total scores are interpreted against validated cutoffs. Cutoff: <26/30 suggests impairment (adjusted for education ≤12 years: +1 point). Total Score: 0-30 (higher = better cognition).
Cognitive changes measured by BACS | 48 hours after last ECT session
  Change in Brief Assessment of Cognition in Schizophrenia (BACS) total score post-treatment.
  BACS is a neuropsychological battery designed to assess cognitive impairment in individuals with schizophrenia. Consists of 6 subtests, each assessing a specific cognitive domain. Raw scores are converted to standardized z-scores (mean = 0, SD = 1) based on normative data. Higher scores = Better cognitive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Psiquiátrico Fray Bernardino Álvarez, México, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting in January 2025
Access Criteria: Access will be granted to researchers who contact the principal investigator directly